CLINICAL TRIAL: NCT02533921
Title: Does Outpatient Palliative Care Improve Patient-centered Outcomes in Parkinson's Disease?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0814
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
Keywords: Palliative Care; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Other): Usual care as in including both a Primary Care Physician (PCP) and neurologist.
  Interventions: Other: Standard of Care
- Interdisciplinary outpatient palliative care (Active Comparator): Usual care augmented by an outpatient interdisciplinary palliative care team.
  Interventions: Other: Interdisciplinary outpatient palliative care

INTERVENTIONS:
Other: Interdisciplinary outpatient palliative care — Interdisciplinary outpatient palliative care is an approach to caring for individuals with life-threatening illnesses that addresses potential causes of suffering including physical symptoms such as pain, psychiatric symptoms such as depression, psychosocial issues and spiritual needs. Palliative care approaches have been successfully applied to improve patient-centered outcomes in cancer as well as several chronic progressive illnesses including heart failure and pulmonary disease.
  Arms: Interdisciplinary outpatient palliative care
Other: Standard of Care — Usual care defined as including both a PCP and neurologist
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to improve outcomes for persons living with Parkinson's Disease (PD) and their family caregivers. The investigators hypothesize that outpatient interdisciplinary palliative care will improve patient-centered outcomes for PD patients at high-risk for poor outcomes.

DETAILED DESCRIPTION:
Palliative care is an approach to caring for individuals with life-threatening illnesses that addresses potential causes of suffering including physical symptoms such as pain, psychiatric symptoms such as depression, psychosocial issues and spiritual needs. Palliative care approaches have been successfully applied to improve patient-centered outcomes in cancer as well as several chronic progressive illnesses including heart failure and pulmonary disease. To date there have been minimal attempts to apply these principles to PD although preliminary evidence suggests that PD patients have significant unmet needs under current models of care which may be amenable through a palliative care model. This study will provide critical information to forward this field including data on the comparative effectiveness of outpatient palliative care for PD versus current standards of care; effects of this intervention on cost and service utilization; and the characteristics of patients most likely to benefit from such an approach and the specific services most needed by PD patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* UK Brain Bank criteria for diagnosis of probable PD or Multiple Systems Atrophy (MSA) or Corticobasal Degeneration (CBD) or Progressive Supranuclear Palsy (PSP) or Lewy Body Dementia (LBD)
* At high risk for poor outcomes as identified by the Palliative Care Needs Assessment Tool (PC-NAT)

Exclusion Criteria:

* Immediate and urgent palliative care needs
* Unable or unwilling to commit to study procedures including;

  1. randomization,
  2. study visits or
  3. the addition of a neurologist to their care team
* Presence of additional chronic medical illnesses which may require palliative services
* Already receiving palliative care and/or hospice services.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09-20 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benzi Kluger, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
- University of Alberta Canada, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Macchi ZA, Miyasaki J, Katz M, Galifianakis N, Sillau S, Kluger BM. Prevalence and Cumulative Incidence of Caregiver-Reported Aggression in Advanced Parkinson Disease and Related Disorders. Neurol Clin Pract. 2021 Dec;11(6):e826-e833. doi: 10.1212/CPJ.0000000000001110. PMID 34992965
- [Derived] Koljack CE, Miyasaki J, Prizer LP, Katz M, Galifianakis N, Sillau SH, Kluger BM. Predictors of Spiritual Well-Being in Family Caregivers for Individuals with Parkinson's Disease. J Palliat Med. 2022 Apr;25(4):606-613. doi: 10.1089/jpm.2020.0797. Epub 2021 Nov 24. PMID 34818097
- [Derived] Kluger BM, Miyasaki J, Katz M, Galifianakis N, Hall K, Pantilat S, Khan R, Friedman C, Cernik W, Goto Y, Long J, Fairclough D, Sillau S, Kutner JS. Comparison of Integrated Outpatient Palliative Care With Standard Care in Patients With Parkinson Disease and Related Disorders: A Randomized Clinical Trial. JAMA Neurol. 2020 May 1;77(5):551-560. doi: 10.1001/jamaneurol.2019.4992. PMID 32040141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Started | 104 | 106
Completed | 88 | 95
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care | Total
Number analyzed (Participants) | 104 | 106 | 210
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data was missing for one person.
  Participants
    number analyzed (Participants) | 103 | 106 | 209
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 19 | 26 | 45
    >=65 years | 84 | 80 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were not available for one participant in the "Standard of Care" Arm
  years
    number analyzed (Participants) | 103 | 106 | 209
    (all) | 70.71 (8.04) | 69.52 (8.25) | 70.11 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 41 | 75
  Male | 70 | 65 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 100 | 103 | 203
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 93 | 100 | 193
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 34 | 67
  United States | 71 | 72 | 143
Presence of Dementia [Count of Participants; unit: Participants] | 30 | 30 | 60
Presence of Caregiver [Count of Participants; unit: Participants] | 88 | 87 | 175
Disease Duration [Mean (Standard Deviation); unit: months] | 114.34 (79.17) | 116.48 (83.70) | 115.42 (81.31)
Quality of Life AD (QOL-AD) [Mean (Standard Deviation); unit: units on a scale] — Higher numbers indicate better outcomes. Scale ranges from 0 to 52.
  units on a scale | 34.29 (5.60) | 33.89 (5.69) | 34.09 (5.64)
Zarit Burden of Care (ZBI) [Mean (Standard Deviation); unit: units on a scale] — Applies only to caregivers. Higher numbers indicate worse outcomes. Scale ranges from 0 to 48.
  units on a scale | 31.27 (8.06) | 32.33 (8.19) | 31.80 (8.12)
Hospital Anxiety and Depression Scale (HADS) - Patient Anxiety [Mean (Standard Deviation); unit: units on a scale] — Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
  units on a scale | 7.73 (4.43) | 7.57 (3.78) | 7.65 (4.11)
Hospital Anxiety and Depression Scale (HADS) - Patient Depression [Mean (Standard Deviation); unit: units on a scale] — Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
  units on a scale | 7.23 (3.74) | 7.04 (3.55) | 7.13 (3.64)
Hospital Anxiety and Depression Scale (HADS) - Caregiver Anxiety [Mean (Standard Deviation); unit: units on a scale] — Only applicable to caregivers. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
  units on a scale | 7.72 (3.57) | 7.14 (3.58) | 7.43 (3.58)
Hospital Anxiety and Depression Scale (HADS) - Caregiver Depression [Mean (Standard Deviation); unit: units on a scale] — Only applicable to caregivers. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
  units on a scale | 4.09 (2.79) | 4.50 (3.34) | 4.30 (3.07)
Montreal Cognitive Assessment (MoCA) Test for Dementia [Mean (Standard Deviation); unit: units on a scale] — Higher numbers indicate better outcomes. Scale ranges from 0 to 30.
  units on a scale | 23.66 (5.08) | 23.96 (4.83) | 23.81 (4.95)
Hoehn and Yar [Count of Participants; unit: Participants] — Higher numbers indicate greater severity of Parkinson's disease.
  Participants
    1 | 0 | 0 | 0
    1.5 | 0 | 2 | 2
    2 | 34 | 25 | 59
    2.5 | 30 | 24 | 54
    3 | 15 | 25 | 40
    4 | 12 | 14 | 26
    5 | 9 | 14 | 23
    Missing | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Subjects Quality of Life (QOL)
Description: The QOL-AD (Quality of Life in Alzheimer's Disease) survey will be used to measure the differences in the quality of life between groups.Higher numbers indicate better outcomes. The scale ranges from 4 to 52.
Time Frame: 0 to 6 months
Population: Available case data for for QOL AD. Longitudinal regression model for all time points. Main outcome is the change from baseline at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 103 | 105
score on a scale | -0.8446 [-1.6807 to -0.00850] | 0.6576 [-0.4299 to 1.7451]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; Comparing the mean within group change from baseline to 6 months between groups. The null hypothesis is there is no mean difference between groups; Test type: Superiority; p = 0.0272, Mixed Models Analysis; Mean Difference (Final Values) = 1.5022, 95% CI 2-sided [0.1706 to 2.8338], Standard Error of Mean 0.6749 — Compares the palliative care plus usual care group to the usual care group

2. Primary Outcome: Changes in Caregiver Distress
Description: The Zarit Caregiver Burden Interview Form (ZBI) will be used to measure differences in Caregiver Distress between groups. Higher scores indicate worse outcomes. Scale ranges from 0 to 48.
Time Frame: 0 to 6 months
Population: Available case data for for ZBI. Applicable only when a caregiver is present. Longitudinal regression model for all time points. Main outcome is the change from baseline at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 87 | 86
score on a scale | -1.2031 [-2.4700 to 0.06381] | -2.3267 [-3.4618 to -1.1917]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1761, Mixed Models Analysis; Mean Difference (Final Values) = -1.1236, 95% CI 2-sided [-2.7569 to 0.5097], Standard Error of Mean 0.8267 — Compares the palliative care plus usual care group to the usual care group

3. Secondary Outcome: Changes in Patient Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to quantify changes in patient anxiety. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
Time Frame: 0 to 6 months
Population: Available case data for for HADS Anxiety. Longitudinal regression model for all time points. Main outcome is the change from baseline at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 102 | 105
score on a scale | -0.7318 [-1.3542 to -0.1094] | -1.1933 [-1.7117 to -0.6750]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2369, Mixed Models Analysis; Mean Difference (Final Values) = -0.4616, 95% CI 2-sided [-1.2291 to 0.3059], Standard Error of Mean 0.3889 — Compares the palliative care plus usual care group to the usual care group

4. Secondary Outcome: Changes in Patient Depression
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to quantify changes in patient depression. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
Time Frame: 0 to 6 months
Population: Available case data for for HADS Depression. Longitudinal regression model for all time points. Main outcome is the change from baseline at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 102 | 105
score on a scale | -0.2041 [-0.7250 to 0.3167] | -0.3351 [-0.9676 to 0.2975]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; Test type: Superiority; p = 0.7484, Mixed Models Analysis; Mean Difference (Final Values) = -0.1309, 95% CI 2-sided [-0.9349 to 0.6730] — Compares the palliative care plus usual care group to the usual care group

5. Secondary Outcome: Changes in Caregiver Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to quantify changes in caregiver anxiety. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
Time Frame: 0 to 6 months
Population: Available case data for for HADS Anxiety for caregiver. Only applicable when a caregiver is present. Longitudinal regression model for all time points. Main outcome is the change from baseline at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 88 | 86
score on a scale | -0.5216 [-1.2056 to 0.1624] | -1.2095 [-1.9032 to -0.5157]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1529, Mixed Models Analysis; Mean Difference (Final Values) = -0.6878, 95% CI 2-sided [-1.6338 to 0.2581], Standard Error of Mean 0.4789 — Compares the palliative care plus usual care group to the usual care group

6. Secondary Outcome: Changes in Caregiver Depression
Description: The Hospital Anxiety and Depression Scale (HADS) will be used to quantify changes in caregiver depression. Higher numbers indicate worse outcomes. Scale ranges from 0 to 21.
Time Frame: 0 to 6 months
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
Number analyzed (Participants) | 88 | 86
score on a scale | -0.1969 [-0.6847 to 0.2910] | -0.3576 [-0.9949 to 0.2797]
Statistical Analysis 1: Comparison: Standard of Care vs Interdisciplinary Outpatient Palliative Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6834, Mixed Models Analysis; Mean Difference (Final Values) = -0.1608, 95% CI 2-sided [-0.9382 to 0.6167], Standard Error of Mean 0.3934 — Compares the palliative care plus usual care group to the usual care group

ADVERSE EVENTS:
Time Frame: 1 year, or for as long as the patient was in the study if they discontinued early.
Description: Coordinators asked patients about common adverse events, including falls and hospitalizations, at every study visit.
Arm/Group | Standard of Care | Interdisciplinary Outpatient Palliative Care
All-Cause Mortality (participants affected / at risk) | 2/104 | 5/106
Serious Adverse Events (participants affected / at risk) | 1/104 | 0/106
Other Adverse Events (participants affected / at risk) | 1/104 | 3/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=104) | Interdisciplinary Outpatient Palliative Care (N=106)
Left proximal humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left femoral head fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=104) | Interdisciplinary Outpatient Palliative Care (N=106)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
substernal pain/ DOE/SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Facial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection secondary to PEG tube insertion (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02533921/Prot_SAP_000.pdf